CLINICAL TRIAL: NCT03985371
Title: An Open-label, Pilot Study to Assess the Safety, Tolerability and Preliminary Efficacy of EDTA Eye Drops on Band Keratopathy
Brief Title: A Pilot Study to Assess the Preliminary Efficacy of EDTA Eye Drops on Band Keratopathy
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Livionex Inc. (Industry)
Responsible Party: Principal Investigator, James V. Aquavella, MD, Professor, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3712
Record Dates: First submitted 2019-06-07; First posted 2019-06-13 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2022-01

CONDITIONS: Corneal Dystrophy, Band-Shaped
Keywords: Band Keratopathy
MeSH Terms: conditions — Corneal Dystrophy, Band-Shaped

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Drops Used (Experimental)
  Interventions: Drug: EDTA Eye Drops

INTERVENTIONS:
Drug: EDTA Eye Drops — One drop in the Band Keratopathy affected eye only, two times per day for six months.

SUMMARY:
The objective of this study is to collect preliminary efficacy and safety data on the use of EDTA EYE Drops (EED) on subjects during an episode of band keratopathy (BK).

DETAILED DESCRIPTION:
This study is an open-label, pilot study of up to 6 subjects with documented BK.

This study has 2 phases: In Phase 1 subjects must be willing to return to the clinic for evaluation of safety and BK symptoms during the treatment period of 6 months (Days 7, 60, 120, 180) and for follow up at Months 9 and 12. In Phase 2 subjects must be willing to return to the clinic at 18 and 24 months post-first dose for a final evaluation.

On Day 1 of the study, potential subjects will be screened and if they meet entry requirements they will be enrolled in the study.

Once enrolled, subjects will be assessed for baseline symptoms and visual acuity, have corneal photographs taken of their affected eye, dispensed EED and instructed to use it for 2 times/day for 6 months in the eye with BK. They will be dosed for the first time in the clinic in order to show them how to consistently use the drops. Subjects will also be given a diary card to record potential adverse events and pain levels (with the first level being noted in the clinic), dismissed from the clinic and reminded to return on Day 7 for assessment of tolerability and safety.

At each subsequent visit (Days 7, 60, 120, 180) the subject will be asked to rate their pain at the time of the visit on a pain analog scale. Their diary card will be reviewed for potential adverse events (AEs) and use of EED will be assessed for technique and compliance. Between visits, subjects will be called every 4 weeks by a member of the study site team to assess potential AEs and dosing compliance.

Additionally, the subject or their caregiver will check the treated eye on a weekly basis and note whether the calcific bands are still present on the diary card. When bands have disappeared, subject will notify the eye clinic and schedule a return visit to obtain corneal photographs and visual acuity test. This may occur outside the planned study visits.

On Day 180, subjects will present at the clinic to return their diary card and unused study product. They will be asked to return to the clinic on Days 270 and 360 for assessment of their visual acuity, pain, corneal photography of the affected eye and potential AEs.

Day 360 will be considered the end of study phase 1. Phase 2 of the study includes long term follow up for possible recurrence. Subjects will be scheduled to return for follow-up visits at months 18 and 24 for assessment of visual acuity and recurrence of BK symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Understand the requirements of the study and provide informed consent prior to undergoing any study-related procedures
2. Be between the ages of 40 and 80 years old, inclusive
3. Have a documented BK diagnosis
4. Be willing and able to comply with protocol-specified dosing, visits to the clinic and tracking of symptoms

Exclusion Criteria:

1. Use other therapies for BK including amniotic membrane or conjunctival grafts.
2. Have other co-morbidities that may confound the safety and efficacy measurements for this study.
3. Have participated in any other clinical trial within 30 days prior to enrollment.
4. Have any condition, abnormality or situation at Baseline that in the opinion of the Principal Investigator may preclude the subject's ability to comply with study requirements, including completion of the study

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-06-29 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Changes of the Cornea | Days 1, 120 and 180 after the start of the study.
  Photographs will be full, direct views taken with a Zeiss model 450 plus split lamp camera.
Change in Snellen Visual Acuity | Days 1, 7, 60, 120 and 180 after the start of the study.
  The Snellen Chart is used to assess visual acuity by asking subjects to read as many of the 11 lines of block letters as they are able.
Change in the Symptoms Associated with Band Keratopathy | Days 1, 7, 60, 180, 270, 360, 540 and 720 after the start of the study.
  Evaluation of pain, as rated by the subject on a visual analog scale, will be the primary symptom assessed throughout this study.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No